CLINICAL TRIAL: NCT06292728
Title: Safety and Feasibility of the ENDOPLY System in Humans: a Pilot Study
Brief Title: ENDOPLY System in Humans: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENDOPLY (Other)
Collaborators: Just 4 Device s.r.o. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ENDOPLY1
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: ENDOPLY System; Endoscopic Gastric Plication; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: ENDOPLY System

INTERVENTIONS:
Device: ENDOPLY System — One endoscopic procedure where the ENDOPLY System is used for endoscopic gastric plication.

SUMMARY:
Prospective, non-randomized study aimed at defining the initial pattern of gastric plication with the ENDOPLY System, and assess feasibility, ergonomics and safety of the device Prospective, single-centre, open label, consecutive enrolment

DETAILED DESCRIPTION:
This is a clinical trial of the ENDOPLY System medical device. Clinical data of 10 obese patients (obesity grade I and II) will be analysed. The ENDOPLY System medical device will be used to perform endoscopic internal plication of the stomach. This clinical trial may lead to an extension of the portfolio of medical devices used to perform endoscopic internal gastric plication.

Participation in this clinical trial may help individual trial subjects follow a strict diet that may lead to weight loss. Weight reduction may improve the overall health, quality of life and life expectancy of the trial subjects, but this cannot be guaranteed.

In this clinical trial, the gastric volume reduction procedure using the ENDOPLY System is performed under general anaesthesia. Under general anaesthesia, the ENDOPLY Platform is inserted through the mouth into the oesophagus and upper stomach, after a preliminary endoscopy for standard evaluation. The 5 mm endoscope allows to choose the initial site of the plications, most likely and according to similar techniques at the incisura (junction between the fundus and the antrum). 10 to 15 ligatures will be placed in the upward directions, thereby narrowing the gastric lumen. The investigator will determine during the procedure if the experimented device suits the regular pattern of plication that have been tested over the years in the literature concerning gastric plication.

Gastric volume reduction procedures using the ENDOPLY System may be associated with risks. There is a possibility of rare or unknown side effects. Risks associated with the investigational device (ENDOPLY System) - expected gastric fold fibrosis without adverse local inflammatory reaction. Patients will be administered standard medications as part of the "Standard of Care" endoscopic gastric examination under general anaesthesia.

Subjects participating in this clinical trial will attend regular follow-up appointments at 1, 3, 6, and 12 months after endoscopic internal plication of the stomach as specified in the study protocol.

ENDOPLY System technical information:

The ENDOPLY medical device does not contain as an integral part a medicinal substance or a derivative of human blood or plasma. The ENDOPLY medical device is not manufactured using tissues of animal origin, in order to minimise the risk of transmission of Transmissible Spongiform Encephalopathy to human. The ENDOPLY medical device complies with the essential the requirements laid down for medical devices in conformity assessment under other legislation governing technical requirements for products, with the exception of those aspects which are the subject of clinical trial. Precautions have been taken to protect health and safety with regard to those aspects of the user and the patients. The ENDOPLY medical device does not have a European Union Certificate for now.

Preliminary tests have included preliminary design-freeze and proof of concept, in-vivo studies at the Veterinary school of Lyon in 3 pigs, with an autopsy at three months and pathology samples analysis that have shown the expected fibrosis of gastric folds without adverse local inflammatory reaction.

ENDOPLY System is made by the company ENDOPLY (Lyon, France). The ENDOPLY System has the same goal as the other devices achieving an internal gastric plication, means APOLLO System (means Apollo Endoscopic surgery), ENDOMINA (means comprised of a triangulation platform and an instrument for tissue piercing and approximation) and Medical's Incisionless Operating Platform-primary obesity surgery endoluminal procedure). The ENDOPLY System aims at narrowing the gastric lumen by the mean of separated folds of the internal gastric wall.

The ENDOPLY Platform - Like its competitors, it is an endoscopic tissue approximation device, with the following parts:

* Handle: it is comprised of two parts that are when the jaws need to be closed.
* The system is made of several channels are put together and assembled within a shaft:
* A 5.6 mm channel for the endoscope (paediatric naso-fibroscope), for the time being.
* A 3 mm channel for the endoscopic grasper.
* A 5 mm channel for the ligature holder.
* The ligature: it consists in a 7 cm plastic barbed special tie made in Polyetheretherketone (PEEK), with a self-adjusting mechanism (locker) and fits into a ligature-holder.
* As a secondary step, a box containing reloads will be installed, thus avoiding frequent in-and-out manipulations. The reload will be also automatized, but those upgrades will not be available for the trial.
* The extremity of the platform, including delivery catheters outside of the inner perimeter (that is out of the patient's mouth), has been designed to be ergonomic.

ELIGIBILITY:
Inclusion Criteria:

1. BMI 30-40, i.e. class I and II obese patients
2. Age above 18 and below 60 years
3. Having failed multiples diet attempts

Exclusion Criteria:

1. Achalasia and other oesophageal motility disorders
2. Severe esophagitis
3. Gastroduodenal ulcer
4. Heart disease and hypertension without treatment
5. Pulmonary, renal or hepatic failure, cancer
6. Pregnancy ongoing, scheduled or in the past months
7. Previous bariatric surgery or endoscopic bariatric technique
8. Participation to another study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time of duration of the ENDOPLY System study procedure | Day 1 - Study Procedure
  Median range of duration of the ENDOPLY System study procedure (hours).
Number of ligatures placed by ENDOPLY System study procedure | Day 1 - Study Procedure
  Mean number of ligatures placed by ENDOPLY System study procedure (mean absolute value)
Gastric perforation events | 12 months
  Number of adverse events related to gastric perforation events (absolute value)
Gastrointestinal bleeding events | 12 months
  Number of adverse event related to gastrointestinal bleeding events (absolute value)
Initial weight-loss | 12 months
  Mean weight loss at timepoints: initial assessment and at 1, 3, 6, 12 months (absolute value of mean weight reduction)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Dargent, MD, Study Director — CEO, chief executive
Locations (1):
- Fakultní nemocnice u sv. Anny v Brně, Gastroenterologické a hepatologické oddělení, Brno, Czechia